CLINICAL TRIAL: NCT06554223
Title: The SUSTAIN 2 Study - SUStained HIV Treatment for Adherence After Interruption in Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ingrid Theresa Katz, M.D., Multiple Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024P001983
Record Dates: First submitted 2024-08-02; First posted 2024-08-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Human Immunodeficiency Virus
Keywords: Differentiated Service Delivery
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUSTAIN-DSD Arm (Experimental): Participants randomized to SUSTAIN-DSD will be enrolled into an Adherence Club and will have 6 months of ART dispensed through a pre-packed dispensing service. Participants may choose to use the decentralized pick-up point solely for medication retrieval or may opt into the peer-support aspect of the Clubs by attending the group session of up to 30 PWH, who will meet once every 6 months in a safe space (e.g., clinic meeting room, church, or local library). At baseline and every 12 months thereafter, a visiting nurse will draw a blood specimen for viral load. Optional process uptake will be recorded. Participants with a raised viral load will be called and offered enhanced adherence counselling; then recalled for a repeat viral load in 3 months.
  Interventions: Behavioral: SUSTAIN-DSD
- Enhanced (guideline-driven) Standard of Care (E-SoC) (Other): As per current SA ART guidelines, all patients who are >28 days late for a scheduled visit are offered enhanced adherence counselling (EAC) at reengagement and restarted on ART. Patients who are >90 days late also have blood drawn for a CD4 count to test for advanced HIV disease. Individual clinic visits occur every 3 months, with 3-month ART dispensing. VL testing is repeated 3 months after restart, then at 12 months and annually there-after, if suppressed. These visits will be managed by clinic staff (nurse or doctor). EAC is a single counselling session delivered by a lay counsellor. The study team will ensure all SoC processes are complete as per the guidelines; and reported to the COCT team as appropriate.
  Interventions: Other: Enhanced (guideline-driven) Standard of Care (E-SoC)

INTERVENTIONS:
Behavioral: SUSTAIN-DSD — Participants randomized to SUSTAIN-DSD will be enrolled into an Adherence Club and will have 6 months of ART dispensed through a pre-packed dispensing service. Participants may choose to use the decentralized pick-up point solely for medication retrieval or may opt into the peer-support aspect of the Clubs by attending the group session of up to 30 PWH, who will meet once every 6 months in a safe space (e.g., clinic meeting room, church, or local library).
  At 6 months, 12 months, and every 12 months thereafter, a visiting nurse will draw a blood specimen for viral load. Optional process uptake will be recorded. Participants with a raised viral load will be called and offered enhanced adherence counselling; then recalled for a repeat viral load in 3 months.
  Arms: SUSTAIN-DSD Arm
Other: Enhanced (guideline-driven) Standard of Care (E-SoC) — As per current SA ART guidelines, all patients who are >28 days late for a scheduled visit are offered enhanced adherence counselling (EAC) at reengagement and restarted on ART. Patients who are >90 days late also have blood drawn for a CD4 count to test for advanced HIV disease. Individual clinic visits occur every 3 months, with 3-month ART dispensing. VL testing is repeated 3 months after restart, then at 12 months and annually there-after, if suppressed.
  These visits will be managed by clinic staff (nurse or doctor). EAC is a single counselling session delivered by a lay counsellor.
  The study team will ensure all SoC processes are complete as per the guidelines; and reported to the COCT team as appropriate.
  Arms: Enhanced (guideline-driven) Standard of Care (E-SoC)

SUMMARY:
The goal of this clinical trial is to learn if the DSD model (SUSTAIN-DSD) is effective in improving participants HIV treatment adherence. The main questions it aims to answer are:

* Does the SUSTAIN-DSD intervention significantly improve participants' treatment adherence and increase rates of viral suppression?
* Does the SUSTAIN-DSD intervention help retain people in care?
* Does SUSTAIN-DSD intervention help reduce the length of treatment interruptions?
* for 24 months, Participants will either receive the SUSTAIN-DSD intervention (i.e. be enrolled in an adherence club where the participants will pick up 6-months of ART medication and have the option to use peer support and additional counseling), and or enhanced standard of care (i.e. visit the clinic for treatment and participate in optional counseling sessions).

Blood will be drawn from the participants at the adherence club visits for viral load tests at baseline and every 12 months.

- Participants will take part in interviews to discuss the participants' experience with the SUSTAIN-DSD intervention.

DETAILED DESCRIPTION:
Differentiated Service Delivery (DSD) models have been shown to provide equivalent or better retention in healthcare and viral (VL) suppression for people with HIV than conventional care models. However, to date, DSD models have been offered only to people with HIV (PWH) considered 'stable' (i.e., retained in care and virally suppressed). Thus, those at high risk of poor outcomes are ineligible for DSD models. In response, the investigators will work with the City of Cape Town to provide the data needed to impact policy guidelines. The investigators designed SUSTAIN2: SUStained HIV Treatment Adherence After INterruption, which will test a scalable, evidence-based DSD model (SUSTAIN-DSD) to address individual, social, and structural barriers to long-term engagement and to increase VL suppression among PWH with an ART treatment interruption or unsuppressed VL (PWH-Gaps).

SUSTAIN-DSD is a six-month adherence club model of care that offers flexible services with multi-month dispensing of medication (de-linked from clinic processes) and support from lay counselors and peers, which has been proven to help PWH to sustain retention and viral suppression in the Western Cape. The study will implement a Hybrid Type 1 randomized controlled trial (RCT) to evaluate the effectiveness of SUSTAIN-DSD on viral suppression among PWH-Gaps at 24 months post-enrollment, as compared to an enhanced standard-of-care (an optimized guidelines-based approach). The investigators will recruit 300 participants from the parent study and clinics (SUSTAIN, R01MH125703, MPI: Orrell/Sabin; UCT Ethics Reference 568/2021), through which the investigators have identified persistent engagement gaps in approximately 45% of the participants, despite adherence counseling, to test this model of care. The investigators will then assess the mechanisms of intervention impact using mixed methods, guided by the Capability, Opportunity, and Motivation model of Behavior (COM-B), and determine implementation outcomes using Proctor's model.

Ultimately, the investigators' goal is to ensure that PWH are able to achieve and maintain virologic suppression through provision of an effective and efficient model of care, which can be used in South Africa's efforts to reach the 2030 goals.

The investigators' central hypothesis is that PWH-Gaps receiving SUSTAIN-DSD will have higher rates of viral suppression than those who receive enhanced routine care. The investigators will use a Hybrid Type 1 RCT design to answer the study questions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years or age)
* Living with HIV
* On a dolutegravir-based first-line ART regimen
* Evidence of a care gap (>28 days late for appointment) or having a raised viral load (≥50 copies/ml) in the preceding year, either from SUSTAIN study data or from clinic records.
* Able to provide full informed consent.
* Willingness to comply with study procedures, including providing regular update of contact details or locator information.

A purposively selected subset of 30 enrolled participants will be invited for a semi-structured, in-depth interview at (or within 2 months after) the month 24 visit (for experience and perceptions; aim 2); and 20 different participants will be invited to participate in in-depth interviews to determine acceptability and feasibility (aim 3) within the same time frame.

Exclusion Criteria at Enrollment:

* Clinical conditions as assessed by the ART clinicians as requiring clinic-based follow-up e.g. tuberculosis or epilepsy.
* Pregnant at enrollment and requiring care in the antenatal clinic system.
* Sustained retention in care (no gaps of >28days) and viral suppression in the preceding year.
* Plans to leave Cape Town permanently within the next 24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Viral suppression (Viral load <50 c/ml) | 24 months post-enrollment
  Viral suppression (Viral load c/ml) will be measured at 24 months post-enrollment.

SECONDARY OUTCOMES:
Viral suppression (Viral load <50 c/ml) at 12 months | 12 months post-enrollment
  Viral suppression (Viral load <50 c/ml) will be measured at 12 months post-enrollment.
Viremia | 12-24 months
  % Plasma VL 50-999 / ≥1000 copies/mL (dichotomous) | Blood Draw and/or NHLS database at 12 and 24 months
Retention in care at study clinics | 12 and 24 months post-enrollment
  Retention in care at study clinics (and in care at any other clinic) will be measured at 12 and 24 months (measured by proportion attending club or clinic visits at months 12 and 24).
Treatment interruptions | 0-24 months post-enrollment
  Treatment interruptions will be measured using pharmacy refill data.
ART adherence using urine tenofovir rapid assays | 12 and 24 months post-enrollment
  ART adherence will be measured using urine tenofovir rapid assays to detect Tenofovir concentrations in participants.
ART adherence using pharmacy data | 12 and 24 months post-enrollment
  ART adherence will be measured using medication possession ratio calculated from pharmacy refill data.
Success in HIV self-management of care | 12 and 24 months post-enrollment
  This outcome will be assessed with the self-regulatory processes 4-item scale, which includes these items:
  I closely monitor whether I take all my ARVs every day (never - always) I make sure that I get new ARVs at the clinic before my ARVs are finished (never - always) If I notice that I have not taken my ARVs or I have taken them too late, I think about what the reason for that was and how I can prevent that from happening again (never - always) I watch carefully that I take all my ARVs every day (never - always)
  Potential responses are given on a scale from 'never' (1) to 'always' (5). The minimum score is 4 and the maximum score is 20. Higher scores are associated with more successful HIV self-management of care.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid T Katz, MD, MHS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified prior to deposit into the repository, but individual-level data will retain a global unique patient identification number to facilitate analyses. The investigators will also make qualitative data available via de-identified transcripts from audio-recorded interviews. The investigators will do so to comply with the NIH requirement that data generated from human subjects be shared broadly. In addition to the subject level data, the investigators will develop and deposit a data dictionary (describing quantitative variables included in datasets), the study protocol, and data collection instruments into the NIMH data archive (NDA) repository to facilitate further analyses and interpretation of data.
Supporting Information: Study Protocol
Time Frame: As required by NDA, the first data submission date will be the second cycle after the grant is awarded, with subsequent submission made bi-annually. Studies will also be created that contain the data used for every publication resulting from the project. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid in findability. The investigators will include that DOI in relevant publications. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now to our knowledge.
Access Criteria: To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.